CLINICAL TRIAL: NCT01165320
Title: A Multicenter, Noncomparative, Open-label Study to Estimate the Safety, Efficacy, and Pharmacokinetics of MK-0991 (Caspofungin) in Japanese Children and Adolescents With Documented Candida or Aspergillus Infections
Brief Title: A Study of Caspofungin (MK-0991) in Japanese Children and Adolescents With Documented Candida or Aspergillus Infections (MK-0991-074)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0991-074; 132240 (Registry Identifier: JAPIC-CTI)
Record Dates: First submitted 2010-07-15; First posted 2010-07-19 (Estimated); Results first posted 2014-04-23 (Estimated); Last update posted 2018-08-27 (Actual); Status verified 2018-07

CONDITIONS: Candidiasis, Esophageal; Candidiasis, Invasive; Aspergillosis
MeSH Terms: conditions — Candidiasis; Candidiasis, Invasive; Aspergillosis | interventions — Caspofungin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Participants with Esophageal Candidiasis (Experimental): Candida infection is strongly suspected based on clinical symptoms and the participant's clinical course, white moss (plaque) is observed on the esophageal mucosa, and therapy via intravenous infusion is judged to be suitable for the present episode of esophageal candidiasis. MK-0991 therapy as a single loading dose of 70 mg/m^2 intravenously on Day 1 (maximum not to exceed 70 mg), followed by 50 mg/m^2 as a single once-daily dose on all subsequent days (maximum of 70 mg daily). The minimum and maximum treatment duration was 7 and 28 days, respectively.
  Interventions: Drug: Caspofungin
- Participants with Invasive Candidiasis (Experimental): Candida infection is strongly suspected based on the presence of refractory fever not responding to an antibiotic agent, or clinical symptoms at the site of disease, or the participant's clinical course. In addition, at least 1 of the following criteria must be met: 1) Candida infection is strongly suspected based on radiographic imaging findings and positive serological test for fungus, 2) yeast is observed by direct microscopy or histopathological test of tissue biopsied from the site of disease, or 3) Candida species are observed by culture test of specimens sampled from the site of disease. MK-0991 therapy as a single loading dose of 70 mg/m^2 intravenously on Day 1 (maximum not to exceed 70 mg), followed by 50 mg/m^2 as a single once-daily dose on all subsequent days (maximum of 70 mg daily). The minimum and maximum treatment duration was 14 and 56 days, respectively.
  Interventions: Drug: Caspofungin
- Participants with Aspergillosis (Experimental): Aspergillus infection is strongly suspected based on clinical symptoms and the participant's clinical course, and characteristic radiographic imaging findings are observed. In addition, at least 1 of the following criteria must be met: 1) risk factors predisposing to an Aspergillus infection, 2) positive serological test for Aspergillus, 3) acute-branching mold with separated hyphae are observed by direct microscopy or histopathological test, or 4) Aspergillus species are observed by culture test. MK-0991 therapy as a single loading dose of 70 mg/m^2 intravenously on Day 1 (maximum not to exceed 70 mg), followed by 50 mg/m^2 as a single once-daily dose on all subsequent days (maximum of 70 mg daily). The minimum and maximum treatment duration was 14 and 84 days, respectively.
  Interventions: Drug: Caspofungin

INTERVENTIONS:
Drug: Caspofungin
  Other Names: MK-0991; CANCIDAS®

SUMMARY:
The study estimates the safety, efficacy, and pharmacokinetics of caspofungin (MK-0991) in Japanese children and adolescents with documented Candida or Aspergillus infections.

ELIGIBILITY:
Inclusion Criteria:

* Japanese patients in whom a causative fungus is detected before treatment with the study drug or patients with strongly suspected deep-seated fungal infection due to Candida species (spp.) or Aspergillus spp.

Exclusion Criteria:

* Patients with mycoses other than ones due to Candida spp. or Aspergillus spp.
* Patients who will receive other systemic antifungal agents for the first time in screening period

Ages: 3 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2010-07-06 (Actual); Primary Completion 2013-09-17 (Actual); Study Completion 2013-09-17 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Mori M, Imaizumi M, Ishiwada N, Kaneko T, Goto H, Kato K, Hara J, Kosaka Y, Koike K, Kawamoto H, Maeda N, Yoshinari T, Kishino H, Takahashi K, Kawahara S, Kartsonis NA, Komada Y. Pharmacokinetics, efficacy, and safety of caspofungin in Japanese pediatric patients with invasive candidiasis and invasive aspergillosis. J Infect Chemother. 2015 Jun;21(6):421-6. doi: 10.1016/j.jiac.2015.01.009. Epub 2015 Jan 30. PMID 25701307
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=0991-074&kw=0991-074&tab=access

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with documented esophageal candidiasis, invasive candidiasis, or aspergillosis and who met all of the additional inclusion and exclusion criteria were to be enrolled in the study
Pre-assignment Details: Three participants were initially enrolled but were withdrawn when their suspected fungal infections were not confirmed. These 3 participants did not receive study drug. No participants with esophageal candidiasis were identified for inclusion in the study.
Groups:
- Participants With Invasive Candidiasis: MK-0991 therapy as a single loading dose of 70 mg/m^2 intravenously on Day 1 (maximum not to exceed 70 mg), followed by 50 mg/m^2 as a single once-daily dose on all subsequent days (maximum of 70 mg daily). The minimum and maximum treatment duration was 14 and 56 days, respectively.
- Participants With Aspergillosis: MK-0991 therapy as a single loading dose of 70 mg/m^2 intravenously on Day 1 (maximum not to exceed 70 mg), followed by 50 mg/m^2 as a single once-daily dose on all subsequent days (maximum of 70 mg daily). The minimum and maximum treatment duration was 14 and 84 days, respectively.
- Participants With Esophageal Candidiasis: MK-0991 therapy as a single loading dose of 70 mg/m^2 intravenously on Day 1 (maximum not to exceed 70 mg), followed by 50 mg/m^2 as a single once-daily dose on all subsequent days (maximum of 70 mg daily). The minimum and maximum treatment duration was 7 and 28 days, respectively.
Period: Overall Study
Arm/Group | Participants With Invasive Candidiasis | Participants With Aspergillosis | Participants With Esophageal Candidiasis
Started | 12 | 8 | 0 (No participants with esophageal candidiasis were identified for inclusion in the study)
Completed | 9 | 4 | 0
Not Completed | 3 | 4 | 0
Not completed — Clinical adverse experience | 2 | 1 | 0
Not completed — Laboratory adverse experience | 1 | 0 | 0
Not completed — Lack of Efficacy | 0 | 2 | 0
Not completed — Reason unknown | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Participants With Invasive Candidiasis | Participants With Aspergillosis | Total
Number analyzed (Participants) | 12 | 8 | 20
Age, Continuous [Mean (Standard Deviation); unit: Years] | 9.8 (5.2) | 9.8 (5.2) | 9.8 (5.0)
Age, Customized [Number; unit: Participants]
  >=3 months and <2 years | 0 | 1 | 1
  >=2 years and <12 years | 8 | 3 | 11
  >=12 years and <18 years | 4 | 4 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 15
  Male | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an Overall Favorable Response to Therapy
Description: Invasive candidiasis: favorable overall response required resolved clinical findings and negative culture test for Candida species on follow-up. If Candida species were not observed in the baseline blood culture, favorable overall response required resolved clinical findings and resolved or improved radiographic findings. Aspergillosis: favorable overall response required resolved, improved, or unchanged clinical findings and resolved or improved radiographic findings, or resolved or improved clinical findings and resolved, improved, or stable radiographic findings.
Time Frame: Invasive candidiasis: up to 56 days; aspergillosis: up to 84 days
Population: The full analysis set included all enrolled participants who received >=1 dose of study drug. No participants with esophageal candidiasis were identified for inclusion in the study and assessment for response to therapy. Participants whose overall response assessment was "unable to judge" were counted as having an unfavorable response.
Measure: Number; unit: Percentage of Participants
Arm/Group | Participants With Invasive Candidiasis | Participants With Aspergillosis
Number analyzed (Participants) | 12 | 8
Percentage of Participants | 66.7 | 62.5

2. Primary Outcome: Percentage of Participants With One or More Drug-Related Adverse Experiences
Description: An adverse experience (AE) is defined as any unfavorable or unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study drug. Any worsening of a preexisting condition which is temporally associated with the use of the study drug is also an AE. A drug-related AE is one judged to be definitely, probably, or possibly related to the study drug.
Time Frame: Invasive candidiasis: up to 70 days; aspergillosis: up to 98 days
Population: The full analysis set included all enrolled participants who received >=1 dose of study drug. No participants with esophageal candidiasis were identified for inclusion in the study and assessment for safety outcomes.
Measure: Number; unit: Percentage of Participants
Arm/Group | Participants With Invasive Candidiasis | Participants With Aspergillosis
Number analyzed (Participants) | 12 | 8
Percentage of Participants | 58.3 | 37.5

ADVERSE EVENTS:
Time Frame: Invasive candidiasis: up to 56 days; aspergillosis: up to 84 days
Description: No participants with esophageal candidiasis were identified for inclusion in the study and assessment for adverse events
Arm/Group | Participants With Invasive Candidiasis | Participants With Aspergillosis
Serious Adverse Events (participants affected / at risk) | 1/12 | 2/8
Other Adverse Events (participants affected / at risk) | 10/12 | 5/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants With Invasive Candidiasis (N=12) | Participants With Aspergillosis (N=8)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants With Invasive Candidiasis (N=12) | Participants With Aspergillosis (N=8)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Bone Marrow Failure (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Ocular Icterus (Eye disorders) | 1 (1) | 0 (0)
Abdominal Discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Hypoaesthesia Oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (4) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0)
Oedema (General disorders) | 1 (1) | 0 (0)
Puncture Site Pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 3 (4) | 0 (0)
Vessel Puncture Site Inflammation (General disorders) | 1 (1) | 0 (0)
Hepatic Function Abnormal (Hepatobiliary disorders) | 2 (2) | 1 (1)
Bacterial Infection (Infections and infestations) | 0 (0) | 1 (1)
Pseudomembranous Colitis (Infections and infestations) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 4 (5) | 1 (1)
Aspartate Aminotransferase Increased (Investigations) | 3 (4) | 1 (1)
Blood Bilirubin Increased (Investigations) | 1 (1) | 0 (0)
Blood Lactate Dehydrogenase Increased (Investigations) | 2 (2) | 0 (0)
Blood Urine Present (Investigations) | 1 (1) | 0 (0)
C-Reactive Protein Increased (Investigations) | 1 (1) | 0 (0)
Gamma-Glutamyltransferase Increased (Investigations) | 3 (3) | 0 (0)
Heart Rate Increased (Investigations) | 0 (0) | 1 (1)
Platelet Count Increased (Investigations) | 1 (1) | 0 (0)
White Blood Cell Count Increased (Investigations) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (3) | 0 (0)
Renal Impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Upper Respiratory Tract Inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 4 (7) | 1 (1)
Angiopathy (Vascular disorders) | 1 (1) | 0 (0)
Venoocclusive Disease (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to publication or presentation. Any information identified by the sponsor as confidential must be deleted prior to submission.